CLINICAL TRIAL: NCT01074996
Title: A Randomized , Open-label, Multicenter, Phase II Study to Compare the Efficacy of S-1 and S-1 Plus Leucovorin as Second Line Treatment on Gemcitabine-refractory Patients With Inoperable or Advanced Pancreatic Cancers
Brief Title: Study of S-1 as Second Line Treatment on Advanced Pancreatic Cancers
Acronym: APC-S1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APC-307PLAH-XJM
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; S-1; S-1 plus Leucovorin; second-line therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination); Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S-1, (Active Comparator): Subjects will receive S-1 until progression
  Interventions: Drug: S-1
- S-1 plus Leucovorin (Experimental): patients will receive S-1 plus Leucovorin until progression
  Interventions: Drug: S-1 plus Leucovorin

INTERVENTIONS:
Drug: S-1 — 40-60mg bid , days 1-14, every 3 weeks
  Arms: S-1,
Drug: S-1 plus Leucovorin — S-1 40-60mg bid, days 1-14 , every 3 weeks Leucovorin 25mg bid , days 1-14 , every 3 weeks
  Arms: S-1 plus Leucovorin

SUMMARY:
A randomized , open-label, multicenter, phase II study to compare the efficacy of S-1 and S-1 plus Leucovorin as second line treatment on gemcitabine-refractory patients with inoperable or advanced pancreatic cancers，investigate the correlation between efficacy and the expressions of thymidylate synthase, dihydropyrimidine dehydrogenase and orotate phosphoribosyltransferase

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed inoperable or APC.
2. Failure of one prior gemcitabine-based regimen was required,chemotherapy used as a radiation sensitizer in the adjuvant or locally advanced setting was not considered as a prior regimen. Patients received last adjuvant gemcitabine-based chemotherapy less than (or equal to) six months can be enrolled into this study.
3. Disease had to be measurable by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
4. Age ≥18 years old.
5. ECOG performance status 0 or 1.
6. Written informed consent and able to comply with the protocol.

Exclusion Criteria:

1. Local (Stage IA to IIB) pancreatic cancer and locally advanced (stage III) pancreatic cancer. Patients relapsing with metastatic disease, after initial diagnoses with local disease can be enrolled into this study.
2. Previous adjuvant radiotherapy for pancreatic cancer, except for patients with progressive lesions outside the radiation port who completed the radiotherapy at least 6 months prior to study entry.
3. More than (or equal to) six months since last adjuvant chemotherapy. Adjuvant therapy without gemcitabine based adjuvant therapy is not allowed. Patient must have recovered from all treatment related toxicity prior to enrollment and must have documented evidence of disease progression (metastatic) following prior chemotherapy.
4. No previous gemcitabine-based therapy for inoperable or APC.
5. Other primary tumour (including primary brain tumours) within the last 5 years prior to enrollment, except for adequately treated carcinoma in situ of the cervix or basal cell skin cancer.
6. Evidence of spinal cord compression or current evidence of central nervous system (CNS) metastases.
7. History or evidence upon neurological exam of CNS disease (unless adequately treated with standard medical therapy) e.g. uncontrolled seizures.
8. Inability to take oral medication, prior surgical procedures affecting absorption or resulting in the requirement for intravenous alimentation or parenteral nutrition with lipids, and/or active peptic ulcer disease
9. Pregnant or lactating females. Serum pregnancy test to be assessed within 7 days prior to study treatment start, or within 14 days with a confirmatory urine pregnancy test within 7 days prior to study treatment start
10. Men and women of childbearing potential (<2 years after last menstruation) not using effective means of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile)
11. Current or recent (within the 30 days prior to starting study treatment) treatment with another investigational drug or participation in another investigational study
12. Evidence of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug, or patient at high risk from treatment complications
13. Known hypersensitivity to any of the study drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-02; Primary Completion 2013-10 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | up to 3 years
  Assuming a 1.8 months median PFS in the S-1 arm, the study was designed to detect an improvement in PFS to 3.5 months in the S-1 plus Leucovorin arm, or 96% prolongation. The calculated number of PFS events needed to detect this difference with α (two-side) of 0.05 and power of 0.8 was 70. Assuming an average enrollment rate of 2.2 patients per month during planned 3-years study period, a total of eighty patients would be able to provide sufficient number of PFS events for the study at end of the study. However, a total of 90 patients were planned for the study, in consideration of comparison for safety and the overall survival between the two treatment groups.

SECONDARY OUTCOMES:
overall survival | up to 3 years
Tumor response rate | up to 3 years
Clinical benefit rate | up to 3 years
safety and tolerance | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xu jianming, M.D., Principal Investigator — The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ge F, Xu N, Bai Y, Ba Y, Zhang Y, Li F, Xu H, Jia R, Wang Y, Lin L, Xu J. S-1 as monotherapy or in combination with leucovorin as second-line treatment in gemcitabine-refractory advanced pancreatic cancer: a randomized, open-label, multicenter, phase II study. Oncologist. 2014 Nov;19(11):1133-4. doi: 10.1634/theoncologist.2014-0223. Epub 2014 Oct 1. PMID 25273077